CLINICAL TRIAL: NCT03084588
Title: Methadone and Interscalene Block for Shoulder Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Glenn Murphy, Director Clinical Research, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EH15-399
Record Dates: First submitted 2016-07-06; First posted 2017-03-21 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Methadone; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methadone (Active Comparator): Patients in the methadone group will receive a single dose of methadone 0.2 mg/kg at induction of anesthesia
  Interventions: Drug: methadone
- Interscalene block (Active Comparator): Patients in the intersclene block group will receive an interscalene block prior to induction of anesthesia
  Interventions: Procedure: Interscalene block

INTERVENTIONS:
Drug: methadone — Patients will be given methadone at induction of anesthesia
  Arms: Methadone
Procedure: Interscalene block — Patients will be given an interscalene block prior to induction of anesthesia
  Other Names: procedure
  Arms: Interscalene block

SUMMARY:
Patients undergoing shoulder surgery may experience moderate-to-severe pain during the first 2-3 days following the operative procedure. Two methods are used to control pain in the early postoperative period. First, an interscalene nerve block (ISB) can be placed prior to surgery to block the pain fibers that supply the shoulder. Although an ISB provides effective analgesia for several hours after surgery, the block is associated with the potential for transient or permanent nerve injury. Furthermore, the ISB can wear off suddenly, resulting in the abrupt onset of severe pain. A second method of pain control involves the use of opioids. Opioids can provide potent pain relief following surgical procedures. However, the agents that are commonly used by anesthesiologists and surgeons only produce pain relief for 2-4 hours, which leads to fluctuations in the levels of pain control. Recent data suggest that the use of a long-acting opioid like methadone in the operating room, which provides analgesia for 24-36 hours, may improve pain control after surgery. The aim of this clinical trial is to compare postoperative pain scores and analgesic requirements in patients randomized to receive either an ISB or methadone at the start of shoulder arthroscopic surgery.

DETAILED DESCRIPTION:
Shoulder surgery is one of the most common orthopedic operations, with 1.4 million procedures performed worldwide. Advances in surgical technology now allow the majority of these procedures to be performed arthroscopically. A growing number of shoulder arthroscopic procedures are now conducted on an outpatient basis. Effective pain control is therefore essential if a patient is to be sent home on the same day as the operation. This management strategy presents an important challenge to anesthesiologists, surgeons, and postanesthesia care unit (PACU) nurses. The pain of a shoulder arthroscopic procedure is equivalent to an open procedure during the first 24-48 hours, and up to 30% of patients report pain of a severe intensity on the first postoperative day. Poor pain control after surgery is associated with lower patient satisfaction scores, adverse events, and the development of chronic postsurgical pain. A variety of therapeutic strategies have been developed to more effectively control this early postoperative pain. However, there are a number of important limitations to each of these approaches.

There are three general approaches that anesthesiologists use to provide anesthesia and analgesia for shoulder arthroscopic surgery. Traditionally, shoulder surgery has been performed with a general anesthetic and a breathing tube (oral endotracheal intubation). Although this provides effective analgesia for the duration of the operation, the patient will experience pain once the intraoperative anesthetic has worn off. In this setting, the anesthesia care provider administers an opioid through the intravenous line so that the patient will awaken in less pain. In the PACU, the nursing staff continues to administer an intravenous opioid until pain is effectively controlled. There are important limitations to this anesthetic management strategy. Anesthesia care providers must estimate the amount of opioid to administer intraoperatively. Since the individual responses to opioids may vary widely, it is possible that patients may awaken in pain or may difficult to extubate (remove the breathing tube) due opioid-induced respiratory depression. Once admitted to the PACU, the patients' pain can be effectively controlled by the careful titration of opioids by nursing staff (pain of less than 3 on a scale of 0 to 10). However, the duration of the effectiveness of commonly-used opioids is only 3-4 hours. Therefore, the patient may have little pain at the time of hospital discharge, but may experience severe pain several hours later. Oral analgesic agents are used to control pain in the home setting. The use of oral opioids results in variability in the level of pain that each patient experiences. This variability is related to the slow onset time and short duration of effect of these oral agents (results in "peaks and troughs" of postoperative pain).

A second anesthetic technique involves the use of a general anesthetic with an interscalene nerve block (ISB). Over 40 years ago, Winnie et al. described the use of a single interscalene brachial plexus block to provide analgesia following shoulder surgery. This practice involves the injection of a large volume of local anesthetic agent near the nerves of the brachial plexus. An ISB or brachial plexus block is a regional anesthetic technique that blocks the nerves that supply the shoulder, arm, and forearm. The block is typically administered in the preoperative holding area before a general anesthetic is performed. When the patient awakens from the general anesthetic and arrives in the PACU, the nerve block provides pain relief which persists for several hours. The risk of nausea and vomiting is also reduced with an ISB block. In addition, most studies have demonstrated that patients randomized to receive an ISB have shorter PACU and hospital length of stays. The advantages of the ISB block have prompted many clinicians to introduce this regional anesthesia technique into their clinical practices. Although an ISB is a very effective postoperative pain management technique, there are several important limitations. The block is usually performed before entering the operating room and may delay the start of the case. In addition, the needle placement for the block is in the neck, and improper placement may result in a pneumothorax (lung collapse). Approximately 5% of ISBs fail, even in experienced hands. Block failure necessitates the use of opioids to control pain. Temporary phrenic nerve palsy or diaphragm paralysis is common after the ISB is performed. This results in a significant decrement in pulmonary function in many patients, including those with normal baseline respiratory muscle strength. Most importantly, clinical investigations, cadaveric studies, and retrospective reviews have suggested that the nerve roots of the brachial plexus may be particularly susceptible to nerve injury from the local anesthetic used for the nerve block. Studies have demonstrated that the ISB is associated with a higher risk of transient and long-term neurologic complications when compared to other peripheral nerve blocks. Furthermore, it is now recognized that the ISB may result in delayed onset phrenic nerve damage and permanent unilateral diaphragmatic paralysis. Finally, the analgesic effects of the ISB may resolve abruptly, resulting in the sudden perception of severe pain. In light of these risks, some experts have questioned the routine use of ISBs for shoulder surgery.

The third strategy for anesthetic and postoperative pain management involves the use an ISB not only as a postoperative analgesic but also as a primary anesthetic. With this approach, an ISB is performed in the preoperative holding area. Once clinicians are assured that the block is functioning, the patient is transported to the operating room, sedation is administered, and the shoulder surgery performed with a combination of sedation and the regional block. Advantages of this technique include the avoidance of general anesthesia (and associated complications), and a better maintenance of blood flow to the brain. A disadvantage of the technique is that a profound nerve block must be present in order for the procedure to be completed successfully. Careful patient selection is also essential when performing shoulder surgery in a sedated patient in the sitting position (anesthesiologists do not have easy access to the patients' airway). Finally, the patient is at risk for all of the complications of ISB listed previously.

When deciding on the appropriate anesthetic for the patient undergoing arthroscopic shoulder surgery, clinicians must weigh the risks and benefits of each technique. As noted above, each anesthetic approach has important limitations. At Evanston hospital, approximately 75% of shoulder surgery patients have an ISB for their procedure. There is a higher utilization of this block at Glenbrook Hospital and at the orthopedic surgery center.

The most important benefit of the ISB is that it provides long-lasting pain relief in the postoperative period. Previous studies have suggested that the analgesic effect of the ISB lasts up to 12 to 24 hours. However, other clinical trials have demonstrated that an ISB provides pain relief for approximately 6 hours, and that pain may be worse after the block has resolved (compared to intravenous opioids). Recently, Abdallah et al. performed a meta-analysis of 23 randomized trials examining 1090 patients to assess the effect of ISBs on pain after shoulder surgery (compared to those not given a block). The authors observed that the duration of pain relief for patients in the ISB group was only 8 hours at rest and 6 hours with movement. There was no further benefit beyond this time. Pain was actually worse at 24 hours in patients given an ISB. These important findings suggest that the effects of the ISB last for a much shorter period of time than estimated by most clinicians, and may impact the evaluation of the risk / benefit ratio of the ISB.

As described previously, an important limitation of the intravenous and oral opioid approach to pain management is that the duration of effect of these agents is only typically 3 to 4 hours. This results in periods of effective pain relief, followed by periods of moderate-to-severe pain in the postoperative period. An alternative strategy for opioid utilization may involve the administration of a very long-acting opioid in the operating room that would provide effective analgesia for the first 24 postoperative hours (which corresponds with the period of the most severe pain after surgery). At the present time, intravenous methadone is the only long-acting opioid available to clinicians. Methadone was developed in 1939 and approved by the FDA for clinical use in 1947. A primary advantage of methadone is its long half-life, which ranges from 25-52 hours when given intravenously in larger doses. This unique property of methadone means that single daily doses can often be used in patients with moderate-to-severe acute or chronic pain. A number of recent investigations have demonstrated that methadone is effective in treating a variety of acute and chronic pain conditions. Although it is best known as a drug used to treat narcotic addiction, methadone is also being used with increasing frequency as an analgesic agent in the operating room to provide prolonged postoperative analgesia. A calculated half-life of 35 hours was observed when methadone was administered intravenously to surgical patients, resulting in a median duration of analgesia lasting 26 hours. In patients undergoing abdominal, orthopedic, cardiac, or gynecologic surgery, the use of a single dose of methadone (20 mg or 0.2-0.3 mg/kg) at induction of anesthesia resulted in improved analgesia for the first 24 hours after surgery, when compared to other intraoperative opioids. In these investigations, patients in the methadone groups required significantly less postoperative pain medication and reported lower pain scores during the first postoperative day. Up to 39% of patients required no additional pain medications, despite undergoing major surgery associated with moderate-to- severe levels of postoperative pain. In a randomized, double-blinded investigation in cardiac surgical patients completed at Evanston Hospital, subjects randomized to the methadone group reported less pain, required reduced postoperative pain medications, and described increased satisfaction with overall pain management when compared to subjects administered a standard opioid (fentanyl). No adverse events directly attributable to methadone were reported in any of these clinical trials.

The use of methadone may be advantageous in the setting of shoulder arthroscopic surgery. The investigators hypothesize that a single dose administered at the start of surgery may provide pain relief throughout the procedure and PACU recovery and for the first 24 hours (or more) after hospital discharge to home. The aim of this clinical trial is to compare analgesia provided by an ISB to that from a pain management strategy using intravenous methadone. Pain scores will be collected from both groups for the first 72 hours after surgery. The requirements for pain medications will also be recorded. Overall satisfaction with pain management will be assessed, and all postoperative complications noted.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting for elective shoulder arthroscopic procedures will be eligible for enrollment.

Exclusion Criteria:

* Preoperative renal failure requiring dialysis
* Poorly controlled pulmonary disease (severe asthma or COPD) -Contraindication to regional anesthesia (recent anticoagulant use)
* Sleep apnea or morbid obesity with possible sleep apnea
* Allergy to methadone
* Significant preoperative pain requiring treatment with high doses of opioids (more than 6-8 Norco tablets or equivalence per day) or recent history of opioid abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-07 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Pain score on a scale of 0 to 10 (0=no pain, 10= worst pain imaginable) | at 24 hours
  scale of 0 to 10 (0=no pain, 10= worst pain imaginable)

SECONDARY OUTCOMES:
Pain score on a scale of 0 to 10 (0=no pain, 10= worst pain imaginable) | at 4 hours after PACU admission
  scale of 0 to 10 (0=no pain, 10 = worst pain imaginable)
hydromorphone consumption | 1 hour after admission
  at PACU dischage
Pain score on a scale of 0 to 10 (0=no pain, 10= worst pain imaginable) | at 48 hours
  scale of 0 to 10 (0=no pain, 10=worst pain imaginable)
Pain score on a scale of 0 to 10 (0=no pain, 10= worst pain imaginable) | at 72 hours
  scale of 0 to 10 (0=no pain, 10=worst pain imaginable)

CONTACTS AND LOCATIONS:
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No